CLINICAL TRIAL: NCT02994836
Title: Anti-TNF Discontinuation in Patients With Inflammatory Bowel Disease: Multicentre, Prospective, Randomized Clinical Trial and Economic Evaluation
Brief Title: GIS-SUSANTI-TNF-2015 (Anti-TNF Discontinuation )
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIS-SUSANTI-TNF-2015
Record Dates: First submitted 2016-10-24; First posted 2016-12-16 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Inflammatory bowel disease; Anti-TNF discontinuation; Ulcerative colitis
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-TNF (Active Comparator): Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use) or Adalimumab (Subcutaneus 40 mg milligram(s)-subcutaneus)
  Interventions: Biological: Anti-TNF: Infliximab (Infusion); Biological: Anti-TNF:Adalimumab (Subcutaneus)
- Anti-TNF discontinuation (Placebo) (Placebo Comparator): Physiological saline solution (Infusion-Intravenous use) or Physiological saline solution (Injection-subcutaneous use)
  Interventions: Drug: Anti-TNF discontinuation: Physiological saline solution

INTERVENTIONS:
Biological: Anti-TNF: Infliximab (Infusion) — Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use)(Visit1,visit 3,visit 4,visit 5, visit 6 and visit 7)
  Arms: Anti-TNF
Drug: Anti-TNF discontinuation: Physiological saline solution — Physiological saline solution (Infusion-Intravenous use)(Visit1,visit 3,visit 4,visit 5, visit 6 and visit 7)
  Arms: Anti-TNF discontinuation (Placebo)
Biological: Anti-TNF:Adalimumab (Subcutaneus) — Adalimumab (Subcutaneus 40 mg milligram(s)-subcutaneus)(Visit 1,visit 2,visit 3,visit 4,visit 5, visit 6 and visit 7).
  Arms: Anti-TNF
Drug: Anti-TNF discontinuation: Physiological saline solution — Physiological saline solution (Injection-subcutaneous use)(Visit 1,visit 2,visit 3,visit 4,visit 5, visit 6 and visit 7).
  Arms: Anti-TNF discontinuation (Placebo)

SUMMARY:
This study will be a multicentre prospective randomized trial to assess the percentage of patients with IBD who, after stopping anti-TNF treatment, have sustained clinical remission at one year compared to those in which the treatment is continued at stable doses

DETAILED DESCRIPTION:
A multicentre prospective randomized trial.

Hypothesis:

The discontinuation of anti-TNF treatment in inflammatory bowel disease (IBD) patients in clinical remission is associated with an increased risk of recurrence compared with maintaining such treatment.

Main objective:

To assess the percentage of patients with IBD who, after stopping anti-TNF treatment, have sustained clinical remission at one year compared to those in which the treatment is continued at stable doses

Secondary objectives:

To compare treatment discontinuation vs. treatment continuation of anti-TNF agents in patients with Crohn´s disease or ulcerative colitis in terms of:

1. remission (relapse-free) time,
2. phenotype changes with both strategies
3. mucosal healing,
4. radiologic healing
5. impact on quality of life and productivity
6. safety
7. to identify relapse predictive factors.
8. To identify relapse predictive factors after anti-TNF drug discontinuation
9. Determining the profile of serum cytokines in patients with both strategies, depending on drug exposure and if maintained clinical remission or relapse.

Planned number of subject to be included: 194

The participation of at 50 hospitals in Spain with an inclusion of about 5 patients per hospital is required..

Case report Form was designed on REDCap (a free, secure, web-based application designed to support data capture for research studies).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBD by the usual criteria; both Crohn's and ulcerative colitis disease.
* Patients older than 18 years.
* In the case of patients with Crohn's disease the indication treatment with anti-TNF it must have been for luminal involvement (no perianal).
* Are currently in clinical remission.
* The clinical remission period with the drug at non-intensified dose it must have been at least 6 months.

The administration of ≥10 mg/kg/8 weeks or 5 mg / kg / ≤ 4 weeks, in the case of infliximab, and 40 mg / week, in the case of adalimumab, is considered an intensified dose.

* At the time of inclusion, the patient should be receiving concomitant immunosuppressants (thiopurine or methotrexate) to anti-TNF treatment, and must have received these immunosuppressive drugs at stable doses for at least the last 3 months.
* In patients with Crohn's disease or ulcerative colitis disease, at baseline colonoscopy (made up to 3 months prior to the screening visit) should not be "significant" injuries.
* In the case of patients with Crohn's ileal or ileocolic disease, in magnetic resonance whole should not be "significant" injuries.(made up to 3 months prior to the screening visit)

Exclusion Criteria:

* Age less than 18 years.
* Patients who have been treated with anti-TNF for other indication than the IBD.
* Patients with Crohn's disease in which the indication for treatment with anti-TNF has been the perianal involvement (or luminal and perianal both); or showing active perianal disease at the time of inclusion.
* Patients who are not receiving concomitant treatment with immunosuppressants (thiopurine or methotrexate) at the moment (and in the previous 3 months).
* Patients undergoing bowel resection surgery; therefore, patients who began anti-TNF therapy to prevent or treat postoperative recurrence in Crohn's disease will be excluded.
* Presence of "significant" endoscopic or radiological lesions
* Advanced chronic illness or any other condition that prevents the patient from coming to the clinic for monitoring or follow-up.
* Patients who are pregnant, breastfeeding or intending to become pregnant during the course of the study.
* Refusal to give consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sustained clinical remission after one year of follow-up (after discontinuing or continuing treatment with anti-TNF). | Change at 12 months.

SECONDARY OUTCOMES:
Clinical activity assessment | Month 0, month 1, month 2, month 4, month 6, month 8, month 10, month 12
  On Crohn´s Disease: Measure by Crohn´s Disease Activity Index (CDAI)
Endoscopic activity assessment | 12 Months. On the Month 0, month 12 or relapse
  On Crohn´s Disease: Measure by Simplified endoscopic activity score for Crohn´s disease (SES-CD).
Radiologic activity assessment | 12 Months. Month 0, month 12 or relapse
  Measure by absence of contrast enhancement, edema or presence of ulcers
Quality of life assessment | Month 0, month 1, month 2, month 4, month 6, month 8, month 10, month 12
  Measure by the Inflammatory Bowel Disease Questionnaire (IBDQ-9)
The Work productivity and activity assessment | Month 0, month 1, month 2, month 4, month 6, month 8, month 10, month 12
  Measure by "Spanish Work Productivity and Activity Impairment Questionnaire".This questionnaire assessments the sum of work time missed because IBD and impairment while working yields the overall work impairment (productivity loss) score. Scores are expressed as percentages of impairment/productivity loss, with higher scores indicating greater impairment.
Clinical activity assessment | Month 0, month 1, month 2, month 4, month 6, month 8, month 10, month 12
  On the Ulcerative Colitis disease: Measure by Mayo Scoring System
Endoscopic activity assessment | 12 Months. On the Month 0, month 12 or relapse
  On the Ulcerative Colitis disease: Measure by Mayo endoscopic score.

CONTACTS AND LOCATIONS:
Overall Officials: Javier MD Perez Gisbert, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

REFERENCES:
- [Background] Lichtenstein GR, Yan S, Bala M, Blank M, Sands BE. Infliximab maintenance treatment reduces hospitalizations, surgeries, and procedures in fistulizing Crohn's disease. Gastroenterology. 2005 Apr;128(4):862-9. doi: 10.1053/j.gastro.2005.01.048. PMID 15825070
- [Background] Clarke K, Regueiro M. Stopping immunomodulators and biologics in inflammatory bowel disease patients in remission. Inflamm Bowel Dis. 2012 Jan;18(1):174-9. doi: 10.1002/ibd.21792. Epub 2011 Jun 14. PMID 21674731
- [Background] Louis E, Belaiche J, Reenaers C. Anti-TNF and Crohn's disease: when should we stop? Curr Drug Targets. 2010 Feb;11(2):148-51. doi: 10.2174/138945010790309957. PMID 20210763
- [Background] Pariente B, Laharie D. Review article: why, when and how to de-escalate therapy in inflammatory bowel diseases. Aliment Pharmacol Ther. 2014 Aug;40(4):338-53. doi: 10.1111/apt.12838. Epub 2014 Jun 23. PMID 24957164
- [Background] Sorrentino D, Nash P, Viladomiu M, Hontecillas R, Bassaganya-Riera J. Stopping anti-TNF agents in patients with Crohn's disease in remission: is it a feasible long-term strategy? Inflamm Bowel Dis. 2014 Apr;20(4):757-66. doi: 10.1097/01.MIB.0000442680.47427.bf. No abstract available. PMID 24572206
- [Background] Solberg IC, Vatn MH, Hoie O, Stray N, Sauar J, Jahnsen J, Moum B, Lygren I; IBSEN Study Group. Clinical course in Crohn's disease: results of a Norwegian population-based ten-year follow-up study. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1430-8. doi: 10.1016/j.cgh.2007.09.002. PMID 18054751
- [Background] Steenholdt C, Molazahi A, Ainsworth MA, Brynskov J, Ostergaard Thomsen O, Seidelin JB. Outcome after discontinuation of infliximab in patients with inflammatory bowel disease in clinical remission: an observational Danish single center study. Scand J Gastroenterol. 2012 May;47(5):518-27. doi: 10.3109/00365521.2012.660541. Epub 2012 Mar 1. PMID 22375898
- [Background] Gisbert JP, Marin AC, Chaparro M. The Risk of Relapse after Anti-TNF Discontinuation in Inflammatory Bowel Disease: Systematic Review and Meta-Analysis. Am J Gastroenterol. 2016 May;111(5):632-47. doi: 10.1038/ajg.2016.54. Epub 2016 Mar 22. PMID 27002797
- [Background] Regueiro M, Kip KE, Baidoo L, Swoger JM, Schraut W. Postoperative therapy with infliximab prevents long-term Crohn's disease recurrence. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1494-502.e1. doi: 10.1016/j.cgh.2013.12.035. Epub 2014 Jan 16. PMID 24440221
- [Background] Bortlík M, Ďuricová D, Lukáš M, Malíčková K, Machková N, Hrdlička L, et al. Infliximab trough levels at treatment discontinuation are associated with increased risk of disease relapse in patients with inflammatory bowel diseases. 20th United European Gastroenterology Week. 2012:P0870.
- [Background] Guidi L, Ratto C, Semeraro S, Roberto I, De Vitis I, Papa A, Marzo M, Parello A, Foglietto G, Doglietto GB, Gasbarrini GB, Fedeli G. Combined therapy with infliximab and seton drainage for perianal fistulizing Crohn's disease with anal endosonographic monitoring: a single-centre experience. Tech Coloproctol. 2008 Jun;12(2):111-7. doi: 10.1007/s10151-008-0411-0. Epub 2008 Jun 10. PMID 18545878
- [Background] Domenech E, Hinojosa J, Nos P, Garcia-Planella E, Cabre E, Bernal I, Gassull MA. Clinical evolution of luminal and perianal Crohn's disease after inducing remission with infliximab: how long should patients be treated? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1107-13. doi: 10.1111/j.1365-2036.2005.02670.x. PMID 16305724
- [Background] Wynands J, Belbouab R, Candon S, Talbotec C, Mougenot JF, Chatenoud L, Schmitz J, Cezard JP, Goulet O, Hugot JP, Ruemmele FM. 12-month follow-up after successful infliximab therapy in pediatric crohn disease. J Pediatr Gastroenterol Nutr. 2008 Mar;46(3):293-8. doi: 10.1097/MPG.0b013e31815604cd. PMID 18376247
- [Background] Dart RJ, Griffin N, Taylor K, Duncan J, Sastrillo M, Sanderson J, Irving PM. Reassessment of Crohn's disease treated with at least 12 months of anti-TNF therapy: how likely is treatment withdrawal? Frontline Gastroenterol. 2014 Jul;5(3):176-182. doi: 10.1136/flgastro-2013-100392. Epub 2013 Dec 24. PMID 28839767
- [Background] Louis E, Mary JY, Vernier-Massouille G, Grimaud JC, Bouhnik Y, Laharie D, Dupas JL, Pillant H, Picon L, Veyrac M, Flamant M, Savoye G, Jian R, Devos M, Porcher R, Paintaud G, Piver E, Colombel JF, Lemann M; Groupe D'etudes Therapeutiques Des Affections Inflammatoires Digestives. Maintenance of remission among patients with Crohn's disease on antimetabolite therapy after infliximab therapy is stopped. Gastroenterology. 2012 Jan;142(1):63-70.e5; quiz e31. doi: 10.1053/j.gastro.2011.09.034. Epub 2011 Sep 22. PMID 21945953
- [Background] Lu C, Waugh A, Bailey RJ, Cherry R, Dieleman LA, Gramlich L, Matic K, Millan M, Kroeker KI, Sadowski D, Teshima CW, Todoruk D, Wong C, Wong K, Fedorak RN. Crohn's disease genotypes of patients in remission vs relapses after infliximab discontinuation. World J Gastroenterol. 2012 Sep 28;18(36):5058-64. doi: 10.3748/wjg.v18.i36.5058. PMID 23049214
- [Background] Molnar T, Lakatos PL, Farkas K, Nagy F, Szepes Z, Miheller P, Horvath G, Papp M, Palatka K, Nyari T, Balint A, Lorinczy K, Wittmann T. Predictors of relapse in patients with Crohn's disease in remission after 1 year of biological therapy. Aliment Pharmacol Ther. 2013 Jan;37(2):225-33. doi: 10.1111/apt.12160. Epub 2012 Nov 26. PMID 23181359
- [Background] Molander P, Farkkila M, Salminen K, Kemppainen H, Blomster T, Koskela R, Jussila A, Rautiainen H, Nissinen M, Haapamaki J, Arkkila P, Nieminen U, Kuisma J, Punkkinen J, Kolho KL, Mustonen H, Sipponen T. Outcome after discontinuation of TNFalpha-blocking therapy in patients with inflammatory bowel disease in deep remission. Inflamm Bowel Dis. 2014 Jun;20(6):1021-8. doi: 10.1097/MIB.0000000000000052. PMID 24798636
- [Background] Echarri A, Ollero V, Gallego C, Porta A, Castro J. Anti-TNF withdrawal in IBD patients on deep remission. Risk factors of relapse. 20th United European Gastroenterology Week. 2012:P0287.
- [Background] Caviglia R, Ribolsi M, Rizzi M, Emerenziani S, Annunziata M, Cicala M. Maintenance of remission with infliximab in inflammatory bowel disease: efficacy and safety long-term follow-up. World J Gastroenterol. 2007 Oct 21;13(39):5238-44. doi: 10.3748/wjg.v13.i39.5238. PMID 17876895
- [Background] Ciria V, Silva P, Leo E, Trigo C, De la Cruz MD, Herrera JM, et al. Factors influencing recurrence following suspension of biological treatment. Importance of mucosal healing. J Crohns Colitis. 2014;8 (suppl.1):P487.
- [Background] Chauvin A, Le Thuaut A, Belhassan M, Le Baleur Y, Mesli F, Bastuji-Garin S, Delchier JC, Amiot A. Infliximab as a bridge to remission maintained by antimetabolite therapy in Crohn's disease: A retrospective study. Dig Liver Dis. 2014 Aug;46(8):695-700. doi: 10.1016/j.dld.2014.04.012. Epub 2014 Jun 2. PMID 24893686
- [Background] Ramos L, Hernandez A, Carrillo M, Alonso I, Hernandez N, Quintero E. Outcome of treatment with biological agents in Crohn's disease: 117 patients in 5 years from a tertiary referral center. J Crohns Colitis. 2014;8 (suppl.1):P398.
- [Background] Luppino I, Spagnuolo R, Marasco R, Cosco C, Ruggiero G, Cosco V, et al. Withdrawal of infliximab (IFX) after achieving remission: outcome in a cohort of inflammatory bowel disease (IBD) patients. Dig Liver Dis. [Conference abstract: Abstracts of the 19th National Congress of Digestive Diseases]. 2013;45S:S100-S1.
- [Background] Marino M, Zucchi E, Fabbro M, Lodolo I, Maieron R, Vadalà S, et al. Outcome of infliximab discontinuation in IBD patients and therapy rechallenging in relapsers: Single centre preliminary data. J Crohns Colitis. 2014;8 (suppl.1):P401.
- [Background] Crombe V, Salleron J, Savoye G, Dupas JL, Vernier-Massouille G, Lerebours E, Cortot A, Merle V, Vasseur F, Turck D, Gower-Rousseau C, Lemann M, Colombel JF, Duhamel A. Long-term outcome of treatment with infliximab in pediatric-onset Crohn's disease: a population-based study. Inflamm Bowel Dis. 2011 Oct;17(10):2144-52. doi: 10.1002/ibd.21615. Epub 2011 Feb 1. PMID 21287665
- [Background] Annunziata ML, Papparella LG, Sansoni I, Balestrieri P, Cicala M. Normalized wall thickness at MRE predicts clinical remission in Crohn's disease after infliximab discontinuation: a 5 years follow-up. J Crohns Colitis. 2014;8 (suppl.1):P402.
- [Background] Waugh AW, Garg S, Matic K, Gramlich L, Wong C, Sadowski DC, Millan M, Bailey R, Todoruk D, Cherry R, Teshima CW, Dieleman L, Fedorak RN. Maintenance of clinical benefit in Crohn's disease patients after discontinuation of infliximab: long-term follow-up of a single centre cohort. Aliment Pharmacol Ther. 2010 Nov;32(9):1129-34. doi: 10.1111/j.1365-2036.2010.04446.x. Epub 2010 Aug 30. PMID 20807218
- [Background] Nuti F, Conte F, Cavallari N, Civitelli F, Aloi M, Alessandri C, et al. Long term efficacy of infliximab in inflammatory bowel disease at a single tertiary center. Dig Liver Dis. [Congress comunication: 17th National Congress SIGENP]. 2010;42(SUPPL. 5):S326-S7.
- [Background] Farkas K, Lakatos PL, Nagy F, Szepes Z, Miheller P, Papp M, Palatka K, Balint A, Bor R, Wittmann T, Molnar T. Predictors of relapse in patients with ulcerative colitis in remission after one-year of infliximab therapy. Scand J Gastroenterol. 2013 Dec;48(12):1394-8. doi: 10.3109/00365521.2013.845906. Epub 2013 Oct 16. PMID 24131338
- [Background] Armuzzi A, Marzo M, Felice C, De Vincentis F, Andrisani G, Moccio G, et al. Long-term scheduled therapy with infliximab in inflammatory bowel disease: a single-centre observational study. Gastroenterology. 2010;238 (suppl.1):S-691.
- [Background] Muñoz C, Bravo MT, Ortiz de Zárate J, Arreba P, García I, Heras J, et al. Mucosal healing in patients with ulcerative colitis treated with infliximab. What happens after treatment is discontinued? J Crohns Colitis. 2014;8 (suppl.1):P405.
- [Background] Dai C, Liu WX, Jiang M, Sun MJ. Mucosal healing did not predict sustained clinical remission in patients with IBD after discontinuation of one-year infliximab therapy. PLoS One. 2014 Oct 20;9(10):e110797. doi: 10.1371/journal.pone.0110797. eCollection 2014. PMID 25330148
- [Background] Casanova MJ, Chaparro M, Garcia-Sanchez V, Nantes O, Leo E, Rojas-Feria M, Jauregui-Amezaga A, Garcia-Lopez S, Huguet JM, Arguelles-Arias F, Aicart M, Marin-Jimenez I, Gomez-Garcia M, Munoz F, Esteve M, Bujanda L, Cortes X, Tosca J, Pineda JR, Manosa M, Llao J, Guardiola J, Perez-Martinez I, Munoz C, Gonzalez-Lama Y, Hinojosa J, Vazquez JM, Martinez-Montiel MP, Rodriguez GE, Pajares R, Garcia-Sepulcre MF, Hernandez-Martinez A, Perez-Calle JL, Beltran B, Busquets D, Ramos L, Bermejo F, Barrio J, Barreiro-de Acosta M, Roncedo O, Calvet X, Hervias D, Gomollon F, Dominguez-Antonaya M, Alcain G, Sicilia B, Duenas C, Gutierrez A, Lorente-Poyatos R, Dominguez M, Khorrami S, Munoz C, Taxonera C, Rodriguez-Perez A, Ponferrada A, Van Domselaar M, Arias-Rivera ML, Merino O, Castro E, Marrero JM, Martin-Arranz M, Botella B, Fernandez-Salazar L, Monfort D, Opio V, Garcia-Herola A, Menacho M, Ramirez-de la Piscina P, Ceballos D, Almela P, Navarro-Llavat M, Robles-Alonso V, Vega-Lopez AB, Moraleja I, Novella MT, Castano-Milla C, Sanchez-Torres A, Benitez JM, Rodriguez C, Castro L, Garrido E, Domenech E, Garcia-Planella E, Gisbert JP. Evolution After Anti-TNF Discontinuation in Patients With Inflammatory Bowel Disease: A Multicenter Long-Term Follow-Up Study. Am J Gastroenterol. 2017 Jan;112(1):120-131. doi: 10.1038/ajg.2016.569. Epub 2016 Dec 13. PMID 27958281
- [Background] Gisbert JP, Panes J. Loss of response and requirement of infliximab dose intensification in Crohn's disease: a review. Am J Gastroenterol. 2009 Mar;104(3):760-7. doi: 10.1038/ajg.2008.88. Epub 2009 Jan 27. PMID 19174781
- [Background] Gisbert JP, Marin AC, Chaparro M. Systematic review: factors associated with relapse of inflammatory bowel disease after discontinuation of anti-TNF therapy. Aliment Pharmacol Ther. 2015 Aug;42(4):391-405. doi: 10.1111/apt.13276. Epub 2015 Jun 15. PMID 26075832
- [Background] Felice C, Pugliese D, Guidi L, Marzo M, Andrisani G, Papa A, et al. Retreatment with infliximab in inflammatory bowel disease: tolerability and effectiveness of different re-induction regimens. J Crohns Colitis. 2014;8 (suppl.1):P363
- [Background] Cabriada JL, Vera I, Domenech E, Barreiro-de Acosta M, Esteve M, Gisbert JP, Panes J, Gomollon F; Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (GETECCU). [Recommendations of the Spanish Working Group on Crohn's Disease and Ulcerative Colitis on the use of anti-tumor necrosis factor drugs in inflammatory bowel disease]. Gastroenterol Hepatol. 2013 Mar;36(3):127-46. doi: 10.1016/j.gastrohep.2013.01.002. Epub 2013 Feb 20. No abstract available. Spanish. PMID 23433780
- [Background] D'Haens G, Feagan B, Colombel JF, Sandborn WJ, Reinisch W, Rutgeerts P, Carbonnel F, Mary JY, Danese S, Fedorak RN, Hanauer S, Lemann M; International Organization for Inflammatory Bowel Diseases (IOIBD) and the Clinical Trial Committee Clincom of the European Crohn's and Colitis Organisation (ECCO). Challenges to the design, execution, and analysis of randomized controlled trials for inflammatory bowel disease. Gastroenterology. 2012 Dec;143(6):1461-9. doi: 10.1053/j.gastro.2012.09.031. Epub 2012 Sep 20. PMID 23000597
- [Background] Daperno M, D'Haens G, Van Assche G, Baert F, Bulois P, Maunoury V, Sostegni R, Rocca R, Pera A, Gevers A, Mary JY, Colombel JF, Rutgeerts P. Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD. Gastrointest Endosc. 2004 Oct;60(4):505-12. doi: 10.1016/s0016-5107(04)01878-4. PMID 15472670
- [Background] Kamm MA, Sandborn WJ, Gassull M, Schreiber S, Jackowski L, Butler T, Lyne A, Stephenson D, Palmen M, Joseph RE. Once-daily, high-concentration MMX mesalamine in active ulcerative colitis. Gastroenterology. 2007 Jan;132(1):66-75; quiz 432-3. doi: 10.1053/j.gastro.2006.10.011. Epub 2006 Oct 12. PMID 17241860
- [Background] Alcala MJ, Casellas F, Fontanet G, Prieto L, Malagelada JR. Shortened questionnaire on quality of life for inflammatory bowel disease. Inflamm Bowel Dis. 2004 Jul;10(4):383-91. doi: 10.1097/00054725-200407000-00009. PMID 15475746
- [Background] Vergara M, Montserrat A, Casellas F, Maudsley M, Gallardo O, Ricart E, Calvet X. Validation of the Spanish Work Productivity and Activity impairment questionnaire: Crohn's disease version. Eur J Gastroenterol Hepatol. 2009 Jul;21(7):809-15. doi: 10.1097/MEG.0b013e32830f4c9e. PMID 19404204
- [Background] Chaparro M, Panes J, Garcia V, Manosa M, Esteve M, Merino O, Andreu M, Gutierrez A, Gomollon F, Cabriada JL, Montoro MA, Mendoza JL, Nos P, Gisbert JP. Long-term durability of infliximab treatment in Crohn's disease and efficacy of dose "escalation" in patients losing response. J Clin Gastroenterol. 2011 Feb;45(2):113-8. doi: 10.1097/MCG.0b013e3181ebaef9. PMID 21242747
- [Background] Brooks AJ, Sebastian S, Cross SS, Robinson K, Warren L, Wright A, Marsh AM, Tsai H, Majeed F, McAlindon ME, Preston C, Hamlin PJ, Lobo AJ. Outcome of elective withdrawal of anti-tumour necrosis factor-alpha therapy in patients with Crohn's disease in established remission. J Crohns Colitis. 2017 Dec 4;11(12):1456-1462. doi: 10.1016/j.crohns.2014.09.007. PMID 25311864
- [Derived] Gisbert JP, Donday MG, Riestra S, Lucendo AJ, Benitez JM, Navarro-Llavat M, Barrio J, Morales-Alvarado VJ, Rivero M, Busquets D, Leo Carnerero E, Merino O, Nantes Castillejo O, Navarro P, Van Domselaar M, Gutierrez A, Alonso-Abreu I, Mejuto R, Fernandez-Salazar L, Iborra M, Martin-Arranz MD, Pineda JR, Sampedro MJ, Serra Nilsson K, Bouhmidi A, Batista L, Munoz Villafranca C, Rodriguez-Lago I, Ceballos D, Guerra I, Manosa M, Marin Jimenez I, Torrella E, Vera Mendoza M, Casanova MJ, de Francisco R, Arias-Gonzalez L, Marin Pedrosa S, Garcia-Bosch O, Garcia-Alonso FJ, Delgado-Guillena P, Garcia MJ, Torrealba L, Nunez-Ortiz A, Vicuna Arregui M, Bosca-Watts MM, Blazquez I, Acosta D, Garre A, Baldan M, Martinez C, Barreiro-de Acosta M, Domenech E, Esteve M, Garcia-Sanchez V, Nos P, Panes J, Chaparro M; EXIT Study group of GETECCU. Withdrawal of antitumour necrosis factor in inflammatory bowel disease patients in remission: a randomised placebo-controlled clinical trial of GETECCU. Gut. 2025 Feb 6;74(3):387-396. doi: 10.1136/gutjnl-2024-333385. PMID 39794921